CLINICAL TRIAL: NCT00298207
Title: Walking Intervention in African American Adults With Newly Diagnosed Hypertension
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Illinois at Chicago (Other)
Responsible Party: Principal Investigator, Augustine J. Sohn, Associate Professor at Department of Family Medicine, University of Illinois at Chicago
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Other
Other Study IDs: 2001-0012
Record Dates: First submitted 2006-02-27; First posted 2006-03-01 (Estimated); Last update posted 2020-03-13 (Actual); Status verified 2020-03

CONDITIONS: Hypertension
Keywords: high blood pressure; hypertension; adult; African Americans; Walking
MeSH Terms: conditions — Hypertension | interventions — Walking

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single Blind

INTERVENTIONS:
Behavioral: Walking (behavior)

SUMMARY:
High blood pressure (hypertension) is one the most common and serious chronic diseases among Americans, especially among the African Americans. The purpose of this study is to explore the effect six month long walking intervention on blood pressure in adult African American with a newly diagnosed high blood pressure (hypertension). The hypothesis is that the group with encouragement to walk extra 30 minutes a day for 5-7 days a week may lower their blood pressure compared to the control group without the encouragement.

DETAILED DESCRIPTION:
Hypertension is a very common and serious chronic disease, which affects approximately 50 million people in the United States. Defined by systolic blood pressure (SBP) of 140 mm Hg or higher or diastolic blood pressure (DBP) of 90 mm Hg or higher, hypertension increases the risk for adverse cardiovascular and renal outcomes, such as myocardial infarction, stroke, congestive heart failure, end-stage renal disease, and peripheral vascular disease. Data from as early as the 1960's indicates that the disease disproportionately effects subgroups of the population, with non-Hispanic African Americans having an age-adjusted prevalence of hypertension (32.4%) almost 40% higher than that noted in non-Hispanic whites (23.3%) and Mexican Americans (22.6%). Although hypertension-related mortality seems to be declining among African Americans, it continues to be a problem which disproportionately affects African Americans more than Whites, particularly in younger age groups.

The management of hypertension is of particular importance for primary care providers, due not only to its prevalence but also because it is a modifiable risk factor for cardiovascular diseases. Although, there are a number of medications available for lowering blood pressure, the first step in managing hypertension should be life-style modification, including weight reduction, increased physical activity, and restriction of dietary sodium and alcohol intake.

Walking seems to be one of the safest and simplest exercises for hypertensive patients of all age groups. Combinations of walking, jogging and bicycling have been shown to be effective in managing hypertension, but there are inherent risks associated with strenuous exercises like jogging and bicycling. Additionally, as most hypertensive patients tend to be overweight, jogging may not be an easy exercise for them. The positive effect of brisk walking on hypertension has been demonstrated in postmenopausal women. Despite the recognized importance of finding ways to effectively manage hypertension in African Americans, there is a paucity of studies on the impact of walking in this population. The purpose of this research was to study the impact of walking an extra 30 minutes a day on blood pressure in 25 to 59 year old African Americans with newly diagnosed hypertension.

ELIGIBILITY:
Inclusion Criteria:

* African American male
* newly diagnosed hypertension
* between age 25 to 59

Exclusion Criteria:

* Not being able to walk unassisted,
* not having telephone access,
* being involved in regular sports activity,
* taking any type of antihypertensive medications,
* advanced renal, cardiovascular, or obstructive pulmonary disease.

Ages: 25 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 20
Dates: Start 2001-04; Study Completion 2004-02

PRIMARY OUTCOMES:
Change in Systolic and diastolic blood pressure over duration of study | Blood Pressure will be measured at study entry, at three months and at six months

CONTACTS AND LOCATIONS:
Overall Officials: Augustine J. Sohn, M.D., M.P.H., Principal Investigator — University of Illinois at Chicago
Locations (1):
- Department of Family Medicine, College of Medicine, University of Illinois at Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Adams PF, Hendershot GE, Marano MA; Centers for Disease Control and Prevention/National Center for Health Statistics. Current estimates from the National Health Interview Survey, 1996. Vital Health Stat 10. 1999 Oct;(200):1-203. PMID 15782448
- [Background] Chobanian AV, Bakris GL, Black HR, Cushman WC, Green LA, Izzo JL Jr, Jones DW, Materson BJ, Oparil S, Wright JT Jr, Roccella EJ; Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. National Heart, Lung, and Blood Institute; National High Blood Pressure Education Program Coordinating Committee. Seventh report of the Joint National Committee on Prevention, Detection, Evaluation, and Treatment of High Blood Pressure. Hypertension. 2003 Dec;42(6):1206-52. doi: 10.1161/01.HYP.0000107251.49515.c2. Epub 2003 Dec 1. PMID 14656957
- [Background] Whelton PK, Perneger TV, Brancati FL, Klag MJ. Epidemiology and prevention of blood pressure-related renal disease. J Hypertens Suppl. 1992 Dec;10(7):S77-84. PMID 1291660
- [Background] Stamler J, Stamler R, Neaton JD. Blood pressure, systolic and diastolic, and cardiovascular risks. US population data. Arch Intern Med. 1993 Mar 8;153(5):598-615. doi: 10.1001/archinte.153.5.598. PMID 8439223
- [Background] Stamler R, Stamler J, Riedlinger WF, Algera G, Roberts RH. Weight and blood pressure. Findings in hypertension screening of 1 million Americans. JAMA. 1978 Oct 6;240(15):1607-10. doi: 10.1001/jama.240.15.1607. PMID 691146
- [Background] Duncan JJ, Farr JE, Upton SJ, Hagan RD, Oglesby ME, Blair SN. The effects of aerobic exercise on plasma catecholamines and blood pressure in patients with mild essential hypertension. JAMA. 1985 Nov 8;254(18):2609-13. PMID 4057469
- [Background] Rogers MW, Probst MM, Gruber JJ, Berger R, Boone JB Jr. Differential effects of exercise training intensity on blood pressure and cardiovascular responses to stress in borderline hypertensive humans. J Hypertens. 1996 Nov;14(11):1369-75. doi: 10.1097/00004872-199611000-00017. PMID 8934367
- [Background] Urata H, Tanabe Y, Kiyonaga A, Ikeda M, Tanaka H, Shindo M, Arakawa K. Antihypertensive and volume-depleting effects of mild exercise on essential hypertension. Hypertension. 1987 Mar;9(3):245-52. doi: 10.1161/01.hyp.9.3.245. PMID 3546120
- [Background] Whelton SP, Chin A, Xin X, He J. Effect of aerobic exercise on blood pressure: a meta-analysis of randomized, controlled trials. Ann Intern Med. 2002 Apr 2;136(7):493-503. doi: 10.7326/0003-4819-136-7-200204020-00006. PMID 11926784
- [Background] Ready AE, Naimark B, Ducas J, Sawatzky JV, Boreskie SL, Drinkwater DT, Oosterveen S. Influence of walking volume on health benefits in women post-menopause. Med Sci Sports Exerc. 1996 Sep;28(9):1097-105. doi: 10.1097/00005768-199609000-00004. PMID 8882996
- [Background] Moreau KL, Degarmo R, Langley J, McMahon C, Howley ET, Bassett DR Jr, Thompson DL. Increasing daily walking lowers blood pressure in postmenopausal women. Med Sci Sports Exerc. 2001 Nov;33(11):1825-31. doi: 10.1097/00005768-200111000-00005. PMID 11689731
- [Background] Lackland DT. Hypertension control among African Americans: an urgent call for action. J Clin Hypertens (Greenwich). 2004 Jun;6(6):333-4. doi: 10.1111/j.1524-6175.2004.03626.x. No abstract available. PMID 15187495
- [Background] Recommendations for routine blood pressure measurement by indirect cuff sphygmomanometry. American Society of Hypertension. Am J Hypertens. 1992 Apr;5(4 Pt 1):207-9. doi: 10.1093/ajh/5.4.207. No abstract available. PMID 1599634
- [Background] Whitt MC, DuBose KD, Ainsworth BE, Tudor-Locke C. Walking patterns in a sample of African American, Native American, and Caucasian women: the cross-cultural activity participation study. Health Educ Behav. 2004 Aug;31(4 Suppl):45S-56S. doi: 10.1177/1090198104266034. PMID 15296691
- [Background] Croteau KA. A preliminary study on the impact of a pedometer-based intervention on daily steps. Am J Health Promot. 2004 Jan-Feb;18(3):217-20. doi: 10.4278/0890-1171-18.3.217. PMID 14748310
- [Background] Iwane M, Arita M, Tomimoto S, Satani O, Matsumoto M, Miyashita K, Nishio I. Walking 10,000 steps/day or more reduces blood pressure and sympathetic nerve activity in mild essential hypertension. Hypertens Res. 2000 Nov;23(6):573-80. doi: 10.1291/hypres.23.573. PMID 11131268
- [Background] Hagburg JM. Exercise, fitness, and hypertension. In: Bouchard C et al., eds. Exercise, Fitness, and Health: A Consensus of Current Knowledge. Champaign, IL: Human Kinetics, 1990. pp. 455-466.
- [Background] Hatano Y. Use of pedometer for promoting daily walking exercise. Int. Council Health Phys Educ Retreat. 1993;29:4-8.